CLINICAL TRIAL: NCT01847118
Title: A Phase Ia, Dose Escalation Study of Humanized Anti-VEGF Monoclonal Antibody (Sevacizumab) Injection in Patients With Advanced or Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM-63-001
Record Dates: First submitted 2013-04-26; First posted 2013-05-06 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2014-07

CONDITIONS: Advanced Solid Tumors; Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sevacizumab (Experimental): 2mg/kg、5mg/kg、7.5mg/kg、10mg/kg、12.5mg/kg、or 15mg/kg. d1, d29, d43, d57
  Interventions: Drug: Sevacizumab

INTERVENTIONS:
Drug: Sevacizumab

SUMMARY:
This study is to assess the safety, tolerability and pharmacokinetics of single dose and multiple doses of humanized anti-VEGF monoclonal antibody (Sevacizumab) in patients with advanced or metastatic solid tumors. The secondary objective is to explore the preliminary anti-tumor effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced or metastatic malignant solid tumors;
* Patients failed the standard anti-tumor therapy or don't have standard regimen;
* At least one measurable lesion;
* At least 4 weeks from the last chemotherapy, 6 weeks from mitomycin, and nitrosourea treatment. If patients received anti-tumor biological products, at least four t1/2 of washout period is needed;
* Toxicity from previous treatment has to restore to ≤ grade 1 (NCI CTC4.0);
* ECOG performance status 0-1;
* Life expectancy ≥ 3 months;
* Adequate hematologic function: ANC ≥ 1.5 × 10^9 /L, HB ≥ 90 g /L (blood transfusion allowed), PLT ≥ 100 × 10^9 /L;
* Adequate hepatic function: ALT ≤ 2.5 × ULN, AST ≤ 2.5 × ULN, TBIL ≤ 1.5 × ULN (patients with liver metastases ALT ≤ 5 × ULN, AST ≤ 5 × ULN, TBIL ≤ 3 × ULN);
* Adequate renal function: creatinine ≤ 1 × ULN;
* Coagulation function: INR ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN;
* Patients of childbearing potential (male and female) must agree to use reliable methods of contraception until at least 12 weeks after the last dose.

Exclusion Criteria:

* HCV, TP or HIV antibody positive;
* Previously received anti-VEGF protein drugs, such as bevacizumab;
* Histologically proven squamous cell lung cancer or squamous cell carcinoma of the head and neck;
* Active hepatitis B infection;
* Evidence of serious infection;
* Symptomatic brain metastases;
* Patients with proteinuria at screening (urine protein ≥ 1+);
* History of abdominal fistula, gastrointestinal perforation, abdominal abscess within 6 months prior to enrollment;
* Serious non-healing wounds, ulcers or fractures;
* Major surgery (excluding biopsy) or significant trauma within 4 weeks prior to enrollment;
* Active bleeding within 3 months prior to enrollment;
* Bleeding diathesis or coagulation disorder;
* History of arterial or venous thrombosis;
* History of myocardial infarction or stroke within 6 months prior to enrollment;
* Unstable angina, congestive heart failure, New York Heart Association (NYHA) class II heart failure, uncontrollable arrhythmia, uncontrolled hypertension (systolic blood pressure> 150 mmHg and/or diastolic blood pressure> 100 mmHg);
* Pregnant and lactating women;
* Known allergies to any excipient in the study drug;
* Patients with alcohol or drug dependence;
* Participation in other clinical trials within 4 weeks before enrollment.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | up to 28 days

SECONDARY OUTCOMES:
Cmax | d1, d2, d5, d8, d11, d15, d18, d22, d25,d29, d43, d57
tmax | d1, d2, d5, d8, d11, d15, d18, d22, d25,d29, d43, d57
AUC | d1, d2, d5, d8, d11, d15, d18, d22, d25,d29, d43, d57
t1/2 | d1, d2, d5, d8, d11, d15, d18, d22, d25,d29, d43, d57
Objective Response Rate (ORR) | d29, d86
Disease Control Rate (DCR) | d29, d86

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China